CLINICAL TRIAL: NCT07058428
Title: Fractionated Stereotactic Radiotherapy Combines With Bevacizumab for the Treatment of Multiple Brain Metastases in Lung Adenocarcinoma: a Prospective Controlled Phase III Study
Brief Title: FSRT Combines With Bevacizumab for Multiple Brain Metastases in Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yet-Sen University Cancer Center (Other)
Responsible Party: Principal Investigator, Hui Liu, chief physician, Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10137
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Multiple Brain Metastases in Lung Adenocarcinoma
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The FSRT+beva group (Experimental): The FSRT+beva group receives FSRT radiotherapy+bevacizumab treatment; FSRT targets visible intracranial lesions with a total dose of 30Gy, administered once a day for a total of 5 times, with a single dose of 6Gy. Bevacizumab starts on day 1 (one week before FSRT treatment), q3w， A total of 4 treatment courses, intravenous injection, with a dose of 7.5mg/kg.
  Interventions: Drug: Bevacizumab; Radiation: FSRT
- The FSRT group (Active Comparator): The FSRT group receives simple FSRT radiotherapy; FSRT is targeted at visible intracranial lesions, with a total dose of 30Gy, administered once a day for a total of 5 days, with a fraction dose of 6Gy.
  Interventions: Radiation: FSRT
- The WBRT group (Active Comparator): The WBRT group receive whole-brain radiotherapy (WBRT) with a simultaneous integrated boost (SIB) to visible intracranial lesions. The prescribed doses are: 40 Gy total to gross lesions and 25 Gy total to the whole brain, delivered in 10 daily fractions.
  Interventions: Radiation: Whole brain radiotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab starts on day 1 (one week before FSRT treatment), q3w，a total of 4 treatment courses, intravenous injection, with a dose of 7.5mg/kg.
  Arms: The FSRT+beva group
Radiation: FSRT — The FSRT group received simple FSRT radiotherapy; FSRT is targeted at visible intracranial lesions, with a total dose of 30Gy, administered once a day for a total of 5 days, with a fraction dose of 6Gy.
  Arms: The FSRT group; The FSRT+beva group
Radiation: Whole brain radiotherapy — The WBRT group received whole brain radiotherapy and locally increased dose radiotherapy for visible intracranial lesions, with a total dose of 40Gy for local lesions and 25Gy for the whole brain, once a day for a total of 10 days.
  Arms: The WBRT group

SUMMARY:
For non-small cell lung cancer brain metastases, stereotactic radiotherapy is gradually replacing whole brain radiotherapy as the standard treatment. When patients have multiple brain metastases or larger tumors (diameter>2cm), single session stereotactic radiotherapy (SRS) may cause significant neurological damage, so fractionated stereotactic radiotherapy (FSRT) is often used. The recent objective remission rate of FSRT is about 50%, and the 1-year intracranial control rate is about 45%, but intracranial progression remains the main factor affecting long-term survival of patients.

Bevacizumab is a recombinant humanized monoclonal antibody against vascular endothelial growth factor, which can improve the efficacy of cranial radiotherapy by normalizing neovascularization and improving the hypoxic state of tumor cells. In addition, bevacizumab can improve the abnormal permeability of neovascularization, reduce exudation and extracellular brain edema, thereby further alleviating the toxic side effects associated with brain radiotherapy.

Based on this, this prospective, controlled phase III study will explore the efficacy and safety of the combined use of fractionated stereotactic radiotherapy and bevacizumab in multiple brain metastases of lung adenocarcinoma.

DETAILED DESCRIPTION:
This prospective, controlled phase III study will explore the efficacy and safety of the combined use of fractionated stereotactic radiotherapy and bevacizumab in multiple brain metastases of lung adenocarcinoma.

Patients will be randomly assigned to three groups in a ratio of 1:1:1. The FSRT+beva group receives FSRT radiotherapy+bevacizumab treatment; FSRT targets visible intracranial lesions with a total dose of 30Gy, administered once a day for a total of 5 days, with a fraction dose of 6Gy. Bevacizumab starts on day 1 (one week before FSRT treatment), q3w， A total of 4 treatment courses, intravenous injection, with a dose of 7.5mg/kg. The FSRT group receives simple FSRT radiotherapy; FSRT is targeted at visible intracranial lesions, with a total dose of 30Gy, administered once a day for a total of 5 days, and a fraction dose of 6Gy for segmentation. The WBRT group receives whole-brain radiotherapy (WBRT) with a simultaneous integrated boost (SIB) to visible intracranial lesions. The prescribed doses are: 40 Gy total to gross lesions and 25 Gy total to the whole brain, delivered in 10 daily fractions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Cellular or histopathological confirmation of lung adenocarcinoma;
* Prior to enrollment, brain enhanced magnetic resonance imaging shows (1) 1-2 brain metastases, with at least one measuring ≥3 cm in diameter; or (2) 3-10 brain metastases, with at least one measuring ≥2 cm in diameter; or (3) 11-20 brain metastases; and deemed unsuitable for single-session SRS by radiation oncologists;
* At the time of enrollment, the extracranial disease status is stable;
* Eastern Cooperative Oncology Group (ECOG) physical fitness status score 0-2 points
* Normal liver, kidney, and bone marrow function within 14 days prior to enrollment: peripheral blood white blood cell count ≥ 4 × 10^9/L; neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, hemoglobin ≥ 100g/L, serum creatinine<1.5 times the upper limit of normal values; Bilirubin<1.5 times the upper limit of normal value; Transaminase<2 times the upper limit of normal value;
* The patient and their family agree and sign an informed consent form.

Exclusion Criteria:

* There are contraindications for bevacizumab, such as a history of cardiac and/or thromboembolic events, or uncontrolled hypertension;
* Meningeal metastasis or extensive intracranial metastasis are not suitable for FSRT;
* Bleeding tendency or coagulation dysfunction;
* Patients with hemoptysis (≥ 1/2 teaspoon of fresh blood per day) within the past month;
* Use full dose anticoagulant therapy within the past month;
* Has experienced severe vascular disease in the past 6 months;
* Have experienced gastrointestinal fistula, perforation, or abdominal abscess within the past 6 months;
* Has experienced hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York Class II or above), acute myocardial infarction, cerebral infarction, cerebral parenchymal hemorrhage, or other active cerebrovascular or cardiovascular diseases within the past 6 months;
* Patients with a history of arterial aneurysm or arteriovenous malformation;
* Having undergone major surgery within 28 days, or minor surgery or needle biopsy within 48 hours;
* Urinary protein 3-4+, or 24-hour urinary protein quantification>1g;
* Simultaneously accompanied by serious and uncontrolled other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression free survival | 2 years
  the time interval from the end of radiotherapy to the first occurrence of intracranial progression or death or the last follow-up;

SECONDARY OUTCOMES:
Progress free survival | 2 years
  Progress free survival (PFS) is defined as the time interval from the end of radiotherapy to the first occurrence of disease progression or death or the last follow-up
Overall survival | 2 years
  Overall survival (OS) is defined as the time interval from the end of radiotherapy to the occurrence of death or the last follow-up
The quality of life (QOL) | 2 years
  The quality of life (QOL) is evaluated using the European Organization for Research and Treatment of Cancer QOL questionnaire version 3.0 (QLQ-C30).
Treatment related side effects | 2 years
  Graded according to CTCAE 5.0
Hopkins Verbal Learning Test-Revised (HVLT-R) Delayed Recall (DR) failure | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
This study is a clinical trial to ensure that patient privacy information is not disclosed.

REFERENCES:
- [Background] Yuan X, Liu WJ, Li B, Shen ZT, Shen JS, Zhu XX. A Bayesian network meta-analysis of whole brain radiotherapy and stereotactic radiotherapy for brain metastasis. Medicine (Baltimore). 2017 Aug;96(34):e7698. doi: 10.1097/MD.0000000000007698. PMID 28834873
- [Background] Boothe D, Young R, Yamada Y, Prager A, Chan T, Beal K. Bevacizumab as a treatment for radiation necrosis of brain metastases post stereotactic radiosurgery. Neuro Oncol. 2013 Sep;15(9):1257-63. doi: 10.1093/neuonc/not085. Epub 2013 Jun 27. PMID 23814264
- [Background] Jiang T, Zhang Y, Li X, Zhao C, Chen X, Su C, Ren S, Yang N, Zhou C. EGFR-TKIs plus bevacizumab demonstrated survival benefit than EGFR-TKIs alone in patients with EGFR-mutant NSCLC and multiple brain metastases. Eur J Cancer. 2019 Nov;121:98-108. doi: 10.1016/j.ejca.2019.08.021. Epub 2019 Sep 27. PMID 31569068
- [Background] Zustovich F, Ferro A, Lombardi G, Zagonel V, Fiduccia P, Farina P. Bevacizumab as front-line treatment of brain metastases from solid tumors: a case series. Anticancer Res. 2013 Sep;33(9):4061-5. PMID 24023350
- [Background] Socinski MA, Langer CJ, Huang JE, Kolb MM, Compton P, Wang L, Akerley W. Safety of bevacizumab in patients with non-small-cell lung cancer and brain metastases. J Clin Oncol. 2009 Nov 1;27(31):5255-61. doi: 10.1200/JCO.2009.22.0616. Epub 2009 Sep 8. PMID 19738122
- [Background] Barrett OC, McDonald AM, Thompson JW, Bredel M, McGwin G, Riley KO, Fiveash JB. Distant brain recurrence in patients with five or more newly diagnosed brain metastases treated with focal stereotactic radiotherapy alone. J Radiosurg SBRT. 2017;4(4):255-263. PMID 28626600
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Mekhail T, Sombeck M, Sollaccio R. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. Curr Oncol Rep. 2011 Aug;13(4):255-8. doi: 10.1007/s11912-011-0180-1. No abstract available. PMID 21584645
- [Background] Baliga S, Garg MK, Fox J, Kalnicki S, Lasala PA, Welch MR, Tome WA, Ohri N. Fractionated stereotactic radiation therapy for brain metastases: a systematic review with tumour control probability modelling. Br J Radiol. 2017 Feb;90(1070):20160666. doi: 10.1259/bjr.20160666. Epub 2016 Dec 12. PMID 27936894
- [Background] Manning MA, Cardinale RM, Benedict SH, Kavanagh BD, Zwicker RD, Amir C, Broaddus WC. Hypofractionated stereotactic radiotherapy as an alternative to radiosurgery for the treatment of patients with brain metastases. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):603-8. doi: 10.1016/s0360-3016(00)00475-2. PMID 10837942
- [Background] Rades D, Janssen S, Dziggel L, Blanck O, Bajrovic A, Veninga T, Schild SE. A matched-pair study comparing whole-brain irradiation alone to radiosurgery or fractionated stereotactic radiotherapy alone in patients irradiated for up to three brain metastases. BMC Cancer. 2017 Jan 6;17(1):30. doi: 10.1186/s12885-016-2989-3. PMID 28061768
- [Background] Serizawa T, Yamamoto M, Higuchi Y, Sato Y, Shuto T, Akabane A, Jokura H, Yomo S, Nagano O, Kawagishi J, Yamanaka K. Local tumor progression treated with Gamma Knife radiosurgery: differences between patients with 2-4 versus 5-10 brain metastases based on an update of a multi-institutional prospective observational study (JLGK0901). J Neurosurg. 2019 Apr 26;132(5):1480-1489. doi: 10.3171/2019.1.JNS183085. Print 2020 May 1. PMID 31026833
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Aoyama H, Tago M, Kato N, Toyoda T, Kenjyo M, Hirota S, Shioura H, Inomata T, Kunieda E, Hayakawa K, Nakagawa K, Kobashi G, Shirato H. Neurocognitive function of patients with brain metastasis who received either whole brain radiotherapy plus stereotactic radiosurgery or radiosurgery alone. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1388-95. doi: 10.1016/j.ijrobp.2007.03.048. PMID 17674975
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Background] Magnuson WJ, Lester-Coll NH, Wu AJ, Yang TJ, Lockney NA, Gerber NK, Beal K, Amini A, Patil T, Kavanagh BD, Camidge DR, Braunstein SE, Boreta LC, Balasubramanian SK, Ahluwalia MS, Rana NG, Attia A, Gettinger SN, Contessa JN, Yu JB, Chiang VL. Management of Brain Metastases in Tyrosine Kinase Inhibitor-Naive Epidermal Growth Factor Receptor-Mutant Non-Small-Cell Lung Cancer: A Retrospective Multi-Institutional Analysis. J Clin Oncol. 2017 Apr 1;35(10):1070-1077. doi: 10.1200/JCO.2016.69.7144. Epub 2017 Jan 23. PMID 28113019
- [Background] Tsao MN, Lloyd N, Wong R, Chow E, Rakovitch E, Laperriere N. Whole brain radiotherapy for the treatment of multiple brain metastases. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD003869. doi: 10.1002/14651858.CD003869.pub2. PMID 16856022
- [Background] Barnholtz-Sloan JS, Sloan AE, Davis FG, Vigneau FD, Lai P, Sawaya RE. Incidence proportions of brain metastases in patients diagnosed (1973 to 2001) in the Metropolitan Detroit Cancer Surveillance System. J Clin Oncol. 2004 Jul 15;22(14):2865-72. doi: 10.1200/JCO.2004.12.149. PMID 15254054
- See also: National Comprehensive Cancer Network. (NCCN) Clinical Practice Guidelines in Oncology. Non-Small Cell Lung Cancer, Version 5. 2019. — https://www.nccn.org/professionals/physician_gls/f_guidelines.asp